CLINICAL TRIAL: NCT06354140
Title: The Efficacy of Tislelizumab Combined With S-1 in Patients With Residual Primary Lesions and Node-Negative Esophageal Squamous Cell Carcinoma After Neoadjuvant Immunochemotherapy Followed by Curative Resection: A Phase II, Multicenter Trial
Brief Title: PPIO-008 Tislelizumab Combined With S-1 in Patients With ypT+N0 ESCC After Radical Resection With Neoadjuvant STUDY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeGuo
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: ypT1-4N0M0
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Tegafur; tislelizumab

STUDY DESIGN:
Masking Description: The study was a one-arm open study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- S-1 Combined With Tislelizumab (Experimental): tegafur (S-1) 80mg/100mg/120mg Q3W (discontinued at the third week) + tislelizumab 200 mg Q3W, treatment for 1 year. tegafur: body surface area (BSA) < 1.25m2, use 80mg; 1.25-1.5m2, use 100mg; > 1.5m2, use 120mg. Treatment for 1 year
  Interventions: Drug: Tegafur

INTERVENTIONS:
Drug: Tegafur — Tegafur (S-1) 80mg/100mg/120mg Q3W (discontinued at the third week) + tislelizumab 200 mg Q3W, treatment for 1 year. Tegafur: body surface area (BSA) < 1.25m2, use 80mg; 1.25-1.5m2, use 100mg; > 1.5m2, use 120mg. Treatment for 1 year
  Other Names: tislelizumab

SUMMARY:
To explore the safety and efficacy of Tegafur combined with tislelizumab in patients with esophageal squamous cell carcinoma with residual primary lesion and node-negative after radical resection following neoadjuvant immunotherapy combined with chemotherapy

DETAILED DESCRIPTION:
Worldwide, esophageal cancer is one of the most common malignancies. According to statistics, the incidence and mortality of esophageal cancer rank 9th and 6th respectively . China is a country with a high incidence of esophageal cancer, with the incidence ranking 6th among all malignant tumors and the mortality ranking 4th among all malignant tumors . The main pathological type of esophageal cancer in China is squamous cell carcinoma, accounting for about 90%. Surgical treatment has always been the main means of esophageal squamous cell carcinoma, but more than 50% of the patients were locally advanced when they were first diagnosed, and the curative effect of simple surgical resection was not ideal. In recent years, the multi-disciplinary integrated treatment mode represented by preoperative induction chemoraotherapy or chemotherapy combined surgery has gradually become the mainstream, and has improved the long-term survival of patients with locally advanced esophageal squamous cell carcinoma to a certain extent. Perioperative comprehensive treatment has gradually become the standard treatment mode for locally advanced esophageal squamous cell carcinoma , and its main comprehensive treatment modes include: 1. Preoperative induction chemotherapy based on the American INT-0113 (RTOG-8911) study , the British OEO2 study and the Japanese JCOG9907 study ; 2. 2. Preoperative induction chemoradiotherapy based on the European CROSS study and the Chinese NEOCRTEC5010 study ; 3. Postoperative adjuvant chemotherapy based on JCOG9204 study .

In spite of the numerous perioperative comprehensive treatment modes, there is still a higher risk of local and distant recurrence and metastasis after the operation of locally advanced esophageal squamous cell carcinoma, and only patients who obtain pathological complete response (pCR) after the preoperative induction therapy may benefit from survival . The pCR rates obtained by preoperative induction chemoradiotherapy reported by different studies were 49% (CROSS study) , 43.2% (NEOCRTEC5010 study) and 33.3% (FFCD9901 study) , respectively. About 50% of the remaining patients (non-PCR) still have a high risk of recurrence and metastasis after surgery. Due to the lack of high-level evidence-based medical evidence, it is controversial whether these patients need complementary adjuvant therapy. For example, clinical guidelines represented by European and American countries only recommend regular follow-up and do not recommend postoperative adjuvant therapy for esophageal squamous cell carcinoma patients who achieve radical resection (R0) regardless of lymph node metastasis. For patients with esophageal adenocarcinoma whose postoperative pathological results indicate positive lymph nodes, supplementary chemotherapy is recommended even for those undergoing radical resection . The clinical guidelines of East Asian countries, represented by Japan, recommend postoperative adjuvant chemotherapy for locally advanced esophageal squamous cell carcinoma with positive lymph nodes confirmed by postoperative pathology. However, for patients with negative lymph nodes after surgery, the CSCO guidelines recommend that for patients who have received neoadjuvant chemoradiotherapy in the past, drug O is recommended as grade II; for patients who have received neoadjuvant chemoradiotherapy, postoperative chemoradiotherapy is recommended as grade III; for patients who have not received neoadjuvant chemoradiotherapy in the past, radiotherapy and chemoradiotherapy are recommended as grade III. At the same time, the postoperative adjuvant of O drug in the NCCN guidelines also requires preoperative radiotherapy and chemotherapy. Therefore, the investigators can see that radiotherapy is required in most cases for postoperative adjuvant therapy of esophageal squamous cell carcinoma. However, for the general clinical and patient compliance considerations in China, the compliance before and after radiotherapy is not high, and the adverse reactions such as esophageal perforation, radiation esophagitis, esophageal obstruction, airway reaction, radiation pneumonia, heart injury and systemic symptoms are likely to occur, which reduces the life treatment and compliance of patients.

In 2020, immunotherapy represented by anti-PD-1 has been established globally in the field of first-line treatment and adjuvant therapy for advanced esophageal cancer and esophagogastric junction cancer. Among them, the results of the CheckMate 649 study showed that first-line treatment with nalizumab combined with chemotherapy (oxaliplatin + fluorouracil regimen) could significantly improve the overall survival (OS) of advanced esophagogastric junction adenocarcinoma patients with PD-L1 comprehensive positive score (CPS ≥ 5) . Similar findings of Attract-4 also suggested that first-line treatment with chemotherapy could improve progression-free survival (PFS) in patients with advanced esophagogastric junction adenocarcinoma, but the benefit of OS was not significant . Keykeynote 590 study results demonstrated that first-line treatment of pabolizumab combined with chemotherapy (cisplatin + fluorouracil regimen) significantly prolonged the survival of advanced esophageal squamous cell carcinoma patients with CPS ≥ 10, although this advantage was not shown in non-selective populations. The results of the CheckMate 577 study are a proof of concept concept) level confirmed that postoperative adjuvant sodium umab can significantly improve the disease-free survival (DFS) of patients with locally advanced esophageal cancer and esophagogastric junction cancer with high risk of recurrence as assessed by pathology after neoadjuvant chemoradiotherapy combined with radical surgery.

According to the results of CheckMate 577, for patients with locally advanced esophageal cancer at or above ypT1 or ypN1 stage after preoperative induction chemoradiotherapy, adjuvant sodium umab therapy could significantly prolong DFS [HR (96.4% CI) 0.69 (0.56 -- 0.86); P = 0.0003]. Although the results of this study have been adopted and recommended by NCCN guidelines as evidence immediately after publication (NCCN 2020 v5.0), the proportion of esophageal squamous cell carcinoma patients is less than 30%, and the patients with postoperative negative lymph nodes have not reached statistical difference, so whether it is consistent with the patient population in China needs further verification. Given the lack of effective adjuvant therapy after surgery for locally advanced esophageal squamous cell carcinoma and the promising preliminary results of PD-1 inhibitors in advanced esophageal squamous cell carcinoma, adjuvant immunotherapy after surgery for esophageal squamous cell carcinoma seems feasible.

As an oral chemotherapy drug, Teggio is more convenient for patients to take. In the study of esophageal cancer, Chen et al. found that CCRT combined with S-1 was tolerable in elderly patients with esophageal cancer, and OS benefited significantly compared with radiotherapy alone. Oral administration of S-1 improves patient compliance, and this regimen is expected to become the preferred regimen for elderly patients with esophageal cancer. Hirahara N et al. studied 20 patients with esophageal squamous cell carcinoma who received neoadjuvant chemotherapy (NAC) and 22 patients who did not receive neoadjuvant chemotherapy during 2011-2020, and took S-1, a one-week rest regimen after 2-week administration, as the tolerance of postoperative adjuvant therapy. One year after surgery, 17 patients (77.2%) in the non-NAC group and 16 patients (80.0%) in the NAC group were still treated with S-1 as planned, and there was no statistically significant difference in the S-1 continuation rate (p = 0.500), indicating that S-1 can be used as a safe and sustainable adjuvant chemotherapy regimen for esophageal cancer patients with or without NAC. Fu et al. included 400 patients treated with postoperative chemotherapy and 582 patients treated with surgery alone. In the chemotherapy group, 69 patients were treated with S-1, 68 with Tegafur tablets, and the rest were treated with intravenous chemotherapy. In the entire study cohort, 3-year OS in the S + CT group was significantly higher than that in the S group (66.3% vs. 49.9%, p < 0.001), these data were confirmed in the matched group (3-year OS, 72.9% vs. 62.0%, p < 0.001). Multivariate Cox regression analysis showed that adjuvant chemotherapy was an independent prognostic factor for ESCC, and patients receiving oral chemotherapy had similar OS as those receiving intravenous chemotherapy. It was also confirmed that adjuvant chemotherapy can significantly improve the OS of pN+ ESCC patients. Compared with intravenous chemotherapy, oral chemotherapy (S-1) has similar efficacy and fewer side effects, which may be a better choice.

For patients with pN0, Wang et al. retrospectively analyzed pT3N0M0 thoracic segment ESCC patients who underwent esophagectomy from January 2008 to December 2012, and used multivariate proportional risk Cox model to determine the factors associated with total recurrence (TR), local recurrence (LR) and distant metastasis (DM). In 692 patients, TR, LR and DM were found to be 35.8% and 41.0%, 28.7% and 32.1%, 16.8% and 21.1%, respectively, at 3 and 5 years, and LR was found to be the main cause of treatment failure in pT3N0M0 thoracic ESCC patients after two fields of dissection. Liu, Zhu et al. [24, 25] all found that the DFS and OS in patients with pN0 treated with postoperative radiotherapy or chemoradiotherapy were significantly higher than those in the group treated with chemotherapy alone, reflecting the effectiveness of adjuvant therapy for pN0 patients.

In summary, the investigators can see that postoperative use of oral oral chemotherapy can bring similar efficacy and better safety to intravenous chemotherapy in patients with pN+ esophageal squamous cell carcinoma. Meanwhile, checkmate577 confirmed that postoperative use of nabriliumab in patients with neoadjuvant chemoratherapy can bring longer DFS in patients with pN+. The adjuvant therapy of postoperative radiotherapy for pN0 patients can also improve the DFS and OS of patients. However, for esophageal squamous cell carcinoma patients who have not received preoperative radiotherapy, the postoperative treatment still needs to be discussed.

Therefore, this project intends to explore the efficacy of postoperative chemtiggio combined with tirellizumab in ESCC patients with esophageal squamous cell carcinoma who have not received neoadjuvant radiotherapy before surgery in patients with radical resection and negative pathological lymph nodes after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Patients with esophageal squamous cell carcinoma with neoadjuvant immunotherapy combined with chemotherapy (radiotherapy was not planned during the study period);
3. Thoracic esophageal squamous cell carcinoma patients with residual pathologic primary site and lymph node positive (ypT1-4aN0M0) after surgery (8th UICC-TNM stage);
4. The operation was radical resection;
5. Physical status ECOG 0 ~ 1 score;
6. No local recurrence or distant metastasis was found in the examination before postoperative adjuvant treatment;
7. There were no contraindications of chemotherapy or immunotherapy in the evaluation of various organ functions;
8. Understand and sign the informed consent.

Exclusion Criteria:

1. Had malignant tumors other than esophageal cancer within 5 years prior to admission (cured localized tumors were not excluded, including cervical carcinoma in situ, skin basal cell carcinoma and prostate carcinoma in situ, etc.); Prostate cancer patients who received hormone therapy and obtained DFS for more than 5 years were not excluded).
2. Prior history of interstitial lung disease, or pneumonia requiring steroid treatment when enrolled;
3. Receiving systemic steroid therapy (more than 10mg of prednisone per day or equivalent) or other immunosuppressant within 2 weeks prior to randomization;
4. People who have been severely allergic to chemotherapy drugs (fluorouracil) or any monoclonal antibody;
5. Patients with active autoimmune diseases;
6. Patients with active hepatitis
7. According to the judgment of the researcher, there are other circumstances that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
1-year DFS rate | Up to 12months
  Rate from surgical resection to local recurrence within one year

SECONDARY OUTCOMES:
Overall survival | Up to 24 months
  From enrollment to death
  From enrollment to death
  From enrollment to death
Progression-free survival | Up to 24 months
  From enrollment to Progression

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No